CLINICAL TRIAL: NCT04583787
Title: xSPECT-based Myocardial Perfusion Scintigraphy: Consistency of Functional Values and Feasibility of Myocardial Uptake Quantitation in Patients With Suspected Coronary Artery Disease (xSPECT MPI Study)
Brief Title: xSPECT-based Myocardial Perfusion Scintigraphy: Consistency of Functional Values and Feasibility of Myocardial Uptake Quantitation in Patients With Suspected Coronary Artery Disease
Acronym: xSPECT MPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Siemens Corporation, Corporate Technology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-02090, qu20Caobelli
Record Dates: First submitted 2020-09-28; First posted 2020-10-12 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Coronary Artery Disease
Keywords: 82Rb-Chloride myocardial perfusion PET with CTCA; 99mTc-sestamibi myocardial perfusion SPECT; Myocardial perfusion SPECT; Absolute myocardial blood flow (MBF); Myocardial Standardized uptake value (SUV); CT coronary angiography (CTCA)
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Patients will receive a 82Rb-PET/CT with CT based coronary angiography (CCTA) as part of clinical care. Subsequently, patients will undergo a stress-rest 99mTc-sestamibi myocardial perfusion SPECT, which will be evaluated both qualitatively and quantitatively
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with suspected CAD (Experimental)
  Interventions: Diagnostic Test: 99mTc-sestamibi myocardial perfusion SPECT; Diagnostic Test: 82Rb-Chloride myocardial perfusion PET with CCTA

INTERVENTIONS:
Diagnostic Test: 99mTc-sestamibi myocardial perfusion SPECT — 82Rb-PET/CT with CT based coronary angiography (CCTA) as part of clinical care at Day 1
Diagnostic Test: 82Rb-Chloride myocardial perfusion PET with CCTA — stress-rest 99mTc-sestamibi myocardial perfusion SPECT, performed subsequent to 99mTc-sestamibi myocardial perfusion SPECT at Day 2

SUMMARY:
This study is to evaluate the feasibility of myocardial Standardized Uptake Volume (SUV) assessment by means of X- (Single photon emission tomography) SPECT/Computed tomography (CT), to assess normal reference value under rest and stress in a homogeneous population without Coronary Artery Disease (CAD) and to assess the variation of absolute quantitative SUV measurements under rest and stress. The values will be evaluated in comparison with perfusion Positron Emission Tomography (PET)/CT (using 82Rb as perfusion tracer) and CT coronary angiography (CTCA) with contrast medium.).

ELIGIBILITY:
Inclusion Criteria:

* Referral to non-invasive nuclear ischemia test as part of clinical care
* Suspected coronary artery disease based on clinical symptoms
* Informed Consent as documented by signature

Exclusion Criteria:

* Pregnancy
* Allergy against adenosine
* Allergy against iodinated contrast medium
* Recent myocardial infarction (<1 month)
* Previous history of coronary revascularization
* Severe asthma
* Thyroid hyperfunction
* atrioventricular block (AV) Block > I grade
* Arrhythmic cardiopathy
* Weight >101 Kg.
* Acute or chronic renal impairment defined as Serum-Creatinine: above 1.5x upper limit of normal (ULN) and/or glomerular filtration rate (GFR) < 30 ml/min
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons,
* Claustrophobia
* Intake of caffeine <24 Hours before the first day of examination
* Enrolment into another study using ionizing radiation within the previous 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Absolute flow quantification (assessed by PET/CT) | 60 minutes at Day 1
  Consistency of quantitative parameters assessed by xSPECT compared to the "gold standard" which includes absolute flow quantification (assessed by PET/CT). The feasibility of myocardial SUV assessment by means of X-SPECT/CT will be tested by correlating the automatically calculated values with automatically calculated, PET-derived absolute blood flows. Rationale: values of quantified myocardial uptake are expected to be reliable the more they correlate with absolutely quantified myocardial blood flow in the myocardium, given the expected proportionality between uptake and subtending coronary blood flow.
presence of significant coronary stenoses (CTCA) | 120 minutes at Day 2
  Consistency of quantitative parameters assessed by xSPECT compared to the "gold standard" which includes the presence of significant coronary stenoses (CTCA). Normal reference values under rest and stress in a homogeneous population without CAD will be evaluated in comparison with perfusion 82Rb-PET/CT and CT coronary angiography (CTCA) with contrast medium. Rationale: a coronary artery disease can be ruled out in patients with normal 82Rb-PET and without detectable stenoses on CTCA, thus identifying a subpopulation of normal patients, wherein reference normal values can be provided.

SECONDARY OUTCOMES:
Determination of uptake patterns that are suggestive for CAD | one point assessment after interventions at day 2
  Values of quantified myocardial uptake (SUV) will be identified and correlated to pathological perfusion patterns as determined by 82Rb-PET/CT.
  Rationale: it is expected that patients with pathological PET imaging and reduced flow rates also present with reduced myocardial uptake of 99mTc-sestamibi.
Quantitative 99mTC-sestamibi uptake values of the whole myocardium | one point assessment after interventions at day 2
  Quantitative 99mTC-sestamibi uptake values of the whole myocardium, analysis of the diagnostic accuracy. Values will be correlated to image-driven diagnosis of CAD Rationale: it is foreseen that a diagnosis can be provided by finding reduced myocardial uptake of 99mTc-sestamibi
Comparison of PET/CT, standard Myocardial perfusion SPECT (MPS) and new quantitative 99mTc-sestamibi xSPECT/quantitative computerized tomography (QCT) in the same patient | one point assessment after interventions at day 2
  Comparison of sensitivity, specificity and accuracy of PET/CT, standard MPS and new quantitative 99mTc-sestamibi xSPECT/QCT in the same patient. Using the final clinical diagnosis of CAD, the diagnostic accuracy of each methodology will be tested by means of receiver operating characteristic (ROC) curves.
  Rationale: it is expected that a quantitative approach can increase the diagnostic accuracy of SPECT by enhancing its sensitivity in case of globally reduced myocardial perfusion, similarly to what gained by quantitative PET
Interobserver variability of all imaging modalities | one point assessment after interventions at day 2
  Interobserver variability of all imaging modalities. A kappa- correlation coefficient will be calculated for all three modalities.
  Rationale: the quantitative data should provide higher interobserver consistency in the evaluation of patients with suspected CAD with SPECT, thus allowing for similar variability compared to quantitative PET.
Interobserver variability of qualitative and quantitative assessments | one point assessment after interventions at day 2
  Interobserver variability of qualitative and quantitative assessments: a kappa correlation coefficient will be evaluated.
  Rationale: the quantitative data should provide higher interobserver consistency in the evaluation of patients with suspected CAD

CONTACTS AND LOCATIONS:
Overall Officials: Federico Caobelli, Dr. med., Principal Investigator — Clinic of Radiology & Nuclear Medicine
Locations (1):
- Clinic of Radiology & Nuclear Medicine, University Hospital of Basel, Basel, Switzerland